CLINICAL TRIAL: NCT05671536
Title: The Effect of Motivational Interviewing Method on Psychological Stability and Treatment Compliance In Hemodialysis Patients
Brief Title: The Effect of Motivational Interview on Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Çiğdem Özdemir Eler, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA21/55
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Hemodialysis
Keywords: Patient on hemodialysis; resilience; nursing; motivational interview
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Patients, undergoing hemodialysis treatment will be assigned to either intervention or control group via simple randomization. Patients on control group will receive standard care. Patients on intervention group will receive 4 sessions of motivational interview at least 20 minutes and once a month. Resilience of all groups will be evaluated at the beginnig of the study and five months after the beginning of the study.
Who Masked: Participant
Masking Description: In order to reduce the selection bias in the determination of intervention and control groups, a list was created by a third party (dialysis center nurse) who did not have a direct role in the study, and intervention and control group assignments were made using the randomization method from the random numbers table. The intervention and control group patients were scheduled to have hemodialysis sessions on different days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview (Experimental): Patients on intervention group will receive 4 sessions of motivational interview at least 20 minutes and once a month. Resilience of patients will be evaluated at the beginnig of the study and five months after the beginning of the study.
  Interventions: Behavioral: motivational interview
- Control (No Intervention): Patients on control group will receive standard care. Resilience of patients will be evaluated at the beginnig of the study and five months after the beginning of the study.

INTERVENTIONS:
Behavioral: motivational interview — Intervention arm will receive motivational interview by the researcher, once a month for 4 times at least 20 minutes. The researcher received education about motivational interview.
  Arms: Motivational interview

SUMMARY:
This research consists of two stages: the first stage aims to evaluate the validity and reliability of the Hemodialysis Resilience Scale, which was developed to evaluate the resilience of patients receiving hemodialysis treatment, in Turkish society, and the second stage aims to determine the effect of motivational interviewing method on patients' psychological resilience and compliance with hemodialysis treatment in individuals undergoing hemodialysis. The main question it aims to answer is:

Does motivational interviewing has an effect on psychological resilience and treatment compliance of hemodialysis patients?

DETAILED DESCRIPTION:
The aims of this study are to evaluate the validity and reliability of the Hemodialysis Resilience Scale, which was developed to evaluate the resilience of patients receiving hemodialysis treatment, in Turkish society, and to determine the effect of motivational interviewing method on patients' psychological resilience and compliance with hemodialysis treatment in individuals undergoing hemodialysis.

This research consists of two stages: the first stage is a methodological study for scale adaptation, and second stage is randomized, controlled, and single blinded study for determining the effect of motivational interviewing.

The first stage is carried out in patients undergoing hemodialysis in two different hospitals. The second stage of the study consists of a randomized, controlled, and single-blinded experimental study to determine the effect of motivational interviewing on individuals undergoing hemodialysis treatment, in terms of psychological resilience and compliance with treatment.

The "simple randomization method" was chosenfor allocation in order to provide an equal number of samples in the two groups. In order to reduce the selection bias in determining intervention and control groups, a list was created by a third party (dialysis center nurse) who did not have a direct role in the study, and assignments were performed using the random numbers table. The intervention and control group patients were scheduled to have hemodialysis sessions on different days. In the study, blinding was applied only to the patient groups because the groups were known by the researchers and nurses.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis treatment for at least 3 months
* 18 years old and over
* Oriantated
* literate
* Having no barrier to written or verbal communication
* Agreed to participate in the research

Exclusion Criteria:

* diagnosed with psychiatric illness
* diagnosed with dementia and Alzheimer's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Resilience | Baseline and 5 months.
  Patient on Hemodialysis Resilience Scale is a valid and 5-point Likert type scale with minimum 0 and maximum 80 points. Higher score means higher resilience. Change=Higher score from Patient on Hemodialysis Resilience Scale at 5 months compared to baseline.
Compliance | Baseline and 5 months.
  End Stage Renal Failure Compliance Scale is a valid and 5-point Likert type scale with minimum 0 and maximum 1200 points. Higher score means higher compliance. Change= Higher score from End Stage Renal Failure Compliance Scale at 5 months compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research will be published after completion and analysis.